CLINICAL TRIAL: NCT04518475
Title: A Multicenter, Randomized, Open-label Study To Compare The Efficacy And Safety Of Eltrombopag Combining Rituximab With Eltrombopag In Adult ITP Patients
Brief Title: Eltrombopag Combining Rituximab Versus Eltrombopag in the Management of Primary Immune Thrombocytopenia (ITP) in Adults
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: The Second Affiliated Hospital of Kunming Medical University (Other); Henan Cancer Hospital (Other Government); Tianjin Medical University Second Hospital (Other); The First Affiliated Hospital of Xiamen University (Other); Nantong University (Other)
Responsible Party: Principal Investigator, Zhang Lei, Professor/Vice director of Thrombosis &Hemostasis Center, Institute of Hematology & Blood Diseases Hospital, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IHBDH-IIT2020014
Record Dates: First submitted 2020-08-12; First posted 2020-08-19 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Primary Immune Thrombocytopenia (ITP)
Keywords: immune thrombocytopenia; autoantibody; eltrombopag; rituximab
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — eltrombopag

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- efficacy of eltrombopag combining rituximab (Experimental): After enrollment,all subjects receive eltrombopag treatment,the initial dose of eltrombopag administration was an oral 75 mg once daily.Complete blood count including platelet count was done once a week.The dose of eltrombopag was adjusted according to the subject platelet count during the period from week 1 to week 24. If the platelet count >250×10^9/L, the eltrombopag will stop until the platelet count <30×10^9/L.
  All subjects receive single dose infusion of rituximab 375 mg/m(2) within 14 days after enrollment.
  Efficacy and safety will be evaluated at Week 4, Week 8, and Week 12.
  Interventions: Drug: eltrombopag combining rituximab
- efficacy of eltrombopag (Active Comparator): After enrollment,all subjects receive eltrombopag treatment,the initial dose of eltrombopag administration was an oral 75 mg once daily.Complete blood count including platelet count was done once a week.The dose of eltrombopag was adjusted according to the subject platelet count during the period from week 1 to week 24. If the platelet count >250×10^9/L, the eltrombopag will stop until the platelet count <30×10^9/L.
  Efficacy and safety will be evaluated at Week 4, Week 8, and Week 12.
  Interventions: Drug: eltrombopag

INTERVENTIONS:
Drug: eltrombopag combining rituximab — After enrollment,all subjects receive eltrombopag treatment,the initial dose of eltrombopag administration was an oral 75 mg once daily.Complete blood count including platelet count was done once a week.The dose of eltrombopag was adjusted according to the subject platelet count during the period from week 1 to week 24. If the platelet count >250×10^9/L, the eltrombopag will stop until the platelet count <30×10^9/L.
  All subjects receive single dose infusion of rituximab 375 mg/m(2) within 14 days after enrollment.
  Efficacy and safety will be evaluated at Week 4, Week 8, and Week 12.
  Other Names: TPO-R agonist & anti-CD20 antibody
  Arms: efficacy of eltrombopag combining rituximab
Drug: eltrombopag — After enrollment,all subjects receive eltrombopag treatment,the initial dose of eltrombopag administration was an oral 75 mg once daily.Complete blood count including platelet count was done once a week.The dose of eltrombopag was adjusted according to the subject platelet count during the period from week 1 to week 24. If the platelet count >250×10^9/L, the eltrombopag will stop until the platelet count <30×10^9/L.
  Efficacy and safety will be evaluated at Week 4, Week 8, and Week 12.
  Other Names: TPO-R agonist
  Arms: efficacy of eltrombopag

SUMMARY:
This multicenter randomized, open-label study aimed to compare the efficacy and safety of eltrombopag combining rituximab with eltrombopag in China adult ITP patients .This study was be conducted in adult ITP patients who had not responded to or had relapsed after previous treatment of ITP, including first line therapy and /or splenectomy.

DETAILED DESCRIPTION:
The primary objective of this study was to evaluate the efficacy and safety of eltrombopag combining rituximab treating previously treated ITP patients compared to eltrombopag. The secondary objective was to evaluate the efficacy of eltrombopag combining rituximab in ITP patients with positive autoantibody compared to eltrombopag .In addition, health-related quality of life (HRQoL) measure was assessed in all participants.

224 eligible subjects were randomized to either eltrombopag combining rituximab or eltrombopag treatment in 1:1 ratio. 112 enrolled patients are randomly picked up to take eltrombopag combining with rituximab at the indicated dose. 112 enrolled patients are randomly picked up to take eltrombopag at the indicated dose.

The initial dose of eltrombopag administration was an oral 75 mg once daily in all participants .The dose of eltrombopag was adjusted according to the subject platelet count during the period from week 1 to week 24.

Subjects in eltrombopag combining rituximab treatment group received single dose infusion of rituximab 375 mg/m(2) within 14 days after enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. Age from 18 to 60 years old
3. Diagnosed with ITP and have a platelet count of <30 ×10^9/L on Day 1 (or within 48 hours prior to dosing on Day 1).
4. Patients who have no response or relapsed after splenectomy(at least more than 6 months). Or patients who have not been splenectomised and have either not responded to one or more prior therapies, or who have relapsed prior therapy.
5. Subjects treated with previous therapy(including but not limited to corticosteroid, azathioprine, danazol, cyclosporin A, mycophenolate mofetil) must have been completed prior to randomization, or must not be increasing a dose after enrollment.
6. No pre-existing cardiac disease within the last 3 months. No arrhythmia known to increase the risk of thrombolic events (e.g. atrial fibrillation), or patients with a Corrected QT interval (QTc) >450msec or QTc >480 for patients with a Bundle Branch Block.
7. No pre-existing infection within the last 1 months(including but not limited to pulmonary infection)
8. Laboratory tests for coagulation function showed that prothrombin time (PT/INR) and activated partial thromboplastin time (APTT) no exceed normal by more than 20%. No history of clotting disorder, other than ITP.
9. White blood cell count, neutrophil absolute value, hemoglobin, within the reference range, with the following exceptions:

   * Hemoglobin: females and males 10.0 g/dl are eligible for inclusion,
   * Absolute neutrophil count (ANC) ≥1500/µL (1.5×109/L) is required for inclusion
10. The following blood chemistry test result no exceed normal by more than 20%:alanine aminotransferase, aspartate aminotransferase, total bilirubin, creatinine,serum albumin must not be below the lower limit of normal (LLN) by more than 10%.
11. Subject is non-childbearing potential of childbearing potential and use acceptable methods of contraception throughout the study.
12. Subjects fully understand and are able to comply with the requirements of the research protocol and are willing to complete the study as planned.

Exclusion Criteria:

1. Patients with any prior history of arterial or venous thrombosis, and with following risk factors: cancer, Factor V Leiden, ATIII deficiency, antiphospholipid syndrome.
2. Pregnant or lactating women;
3. Subjects is currently receiving treatment with another study medication.
4. Any laboratory or clinical evidence for HIV infection.
5. Any clinical history for hepatitis C infection; chronic hepatitis B infection; or any evidence for active hepatitis at the time of subject screening. Laboratory test shows positive serology for Hepatitis C or Hepatitis B (HB). In addition, if negative for HBsAg but HBcAb positive (regardless of HBsAb status), a HB DNA test will be performed and if positive the subject will be excluded.
6. History of platelet aggregation that prevents reliable measurement of platelet counts.
7. Any clinically relevant abnormality, other than ITP,which in the opinion of the investigator makes the subject unsuitable for participation in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 224 (Estimated)
Dates: Start 2020-08-10 (Actual); Primary Completion 2022-02-10 (Estimated); Study Completion 2022-08-10 (Estimated)

PRIMARY OUTCOMES:
Treatment response | From the start of study treatment (Day 1) up to the end of week 12.
  Number of participants achieving a platelet count >=30×10^9/L and at least doubling of the baseline count at Week 4, Week 8, and Week 12 .

SECONDARY OUTCOMES:
Drug efficacy | From the start of study treatment (Day 1) up to the end of week 4, week 8 and week 12.
  Number of participants achieving a platelet count >=30×10^9/L at week 4, week 8, and week 12 in ITP patients with positive autoantibody
Long-term treatment response | From the start of study treatment (Day 1) up to the end of week 16, week 20 and week 24
  Number of participants achieving a platelet count >=30×10^9/L at week 16, week 20, and week 24.
Time to Response | From the start of study treatment (Day 1) up to the end of week 24
  Time to response is defined as time from the start of treatment to the first time of achieving a platelet count >=30×10^9/L and at least doubling of the baseline count during the whole 24 weeks.
Duration of response | From the start of study treatment (Day 1) up to the end of week 24.
  Total duration of time a participant had a platelet count >=30×10^9/L
Evaluation of effectiveness | From the start of study treatment (Day 1) up to the end of week 24.
  Number of participants that reduced or discontinued baseline concomitant ITP medications during the whole 24 weeks.
Number of participants with clinically significant bleeding as assessed using the world health organization (WHO) bleeding scale. | From the start of study treatment (Day 1) up to the end of week 24.
  The WHO Bleeding Scale is a measure of bleeding severity with the following grades: grade 0 = no bleeding, grade 1= petechiae, grade 2= mild blood loss, grade 3 = gross blood loss, and grade 4 = debilitating blood loss.
Immune Thrombocytopenia Patient Assessment Questionnaire (ITP-PAQ) | From the start of study treatment (Day 1) up to the end of week 24.
  In all participants ,use ITP-PAQ to assess the HRQoL before and after treatment.
Functional Assessment of Chronic Illness Therapy fatigue subscale (FACIT-F) | From the start of study treatment (Day 1) up to the end of week 24.
  In all participants ,use FACIT-F to assess the HRQoL before and after treatment.
Number of Participants with side effects of the drugs | From the start of study treatment (Day 1) up to the end of week 24.
  Side effects of the drugs included fever, headache, serum disease,hypotension, rashes, infection liver injury, hypokalaemia, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, M.D., Ph.D, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Institute of Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Tianjin, China

IPD SHARING:
Plan to Share IPD: No